CLINICAL TRIAL: NCT03353012
Title: Acceptability & Tolerance of Immediate Versus Delayed Postpartum Contraceptive Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sitanan Lertsiripanich
Record Dates: First submitted 2017-10-15; First posted 2017-11-24 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2017-10

CONDITIONS: Breastfeeding; Post Partum
Keywords: Immediate postpartum implant; postpartum implant; implant contraception; Etonogestrel; Levonorgestrel
MeSH Terms: conditions — Breast Feeding | interventions — etonogestrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Levonorgestrel immediate post-partum (Experimental): Breast-feeding postpartum woman who receive Levonorgestrel drug implant (75 mg) between 48-72 hr after child delivery
  Interventions: Drug: Levonorgestrel Drug Implant
- Etonogestrel immediate post-partum (Experimental): Breast-feeding postpartum woman who receive Etonogestrel drug implant (68 mg) between 48-72 hr after child delivery
  Interventions: Drug: Etonogestrel Drug Implant
- Levonorgestrel delayed post-partum (Active Comparator): Breast-feeding postpartum woman who receive Levonorgestrel drug implant (75 mg) between 5-7 weeks after child delivery
  Interventions: Drug: Levonorgestrel Drug Implant
- Etonogestrel delayed post-partum (Active Comparator): Breast-feeding postpartum woman who receive Etonogestrel drug implant (68 mg) between 5-7 weeks after child delivery
  Interventions: Drug: Etonogestrel Drug Implant

INTERVENTIONS:
Drug: Etonogestrel Drug Implant — Etonogestrel 68 mg (single rod) is implanted at inner arm of participant.
  Other Names: Implanon
  Arms: Etonogestrel delayed post-partum; Etonogestrel immediate post-partum
Drug: Levonorgestrel Drug Implant — Levonorgestrel 75 mg (2 rods) are implanted at inner arm of participant.
  Other Names: Jadelle
  Arms: Levonorgestrel delayed post-partum; Levonorgestrel immediate post-partum

SUMMARY:
To study and compare acceptability and tolerance between breast-feeding post-partum woman, who receive contraceptive implant 48-72 hours after giving birth or at 5-7 weeks after giving birth, using either Levonorgestrel or Etonogestrel contraceptive implant.

DETAILED DESCRIPTION:
* To study and compare acceptability and tolerance between breast-feeding post-partum woman, who receive contraceptive implant 48-72 hours after giving birth or at 5-7 weeks after giving birth, using either Levonorgestrel or Etonogestrel contraceptive implant.
* Participants who wish to attend the study will be invited to choose between Levonorgestrel and Etonogestrel contraceptive implant, then they will be randomized into immediate postpartum or delay postpartum group. They will be follow-up at 6 and 12 weeks after receive contraceptive implant.
* Information about side effects, breastfeeding status, child growth, acceptability and tolerance will be noted using medical records and interviewing, gathering on paper case record forms.
* Sample size N = 60 (30 in each group (Immediate and delay postpartum group, 15 in each subgroup (Levonogestrel and Etonogestrel group)) This number of sample size is already counted with 10% data loss

ELIGIBILITY:
Inclusion Criteria:

* Breast-feeding post-partum woman aged 18-45 years who wish to use contraceptive implant

Exclusion Criteria:

* Pregnant
* Woman who has any medical conditions which is considered contraindicated to use contraceptive implant
* Woman with severe antepartum or peripartum complications
* Woman who is contraindicated to breastfeed.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | immediately after contraceptive implant use until 12 weeks after use
  To compare treatment-related adverse events between Immediate and delayed breastfeeding postpartum contraceptive users, using case record form which specify bleeding days, spotting days, abdominal discomfort, headache, acne, alopecia, weight and blood pressure of users.
Removal rate of contraceptive implants users | immediately after contraceptive implant use until 12 weeks after use
  To compare tolerance between Immediate and delayed breastfeeding postpartum contraceptive users, by collecting and calculating removal rate of users.
Satisfactory of contraceptive implant users | immediately after contraceptive implant use until 12 weeks after use
  To compare acceptability between Immediate and delayed breastfeeding postpartum contraceptive users, using questionnaire rating satisfactory scale by score from 1 to 5

SECONDARY OUTCOMES:
Breastfeeding status | immediately after contraceptive implant use until 12 weeks after use
  To compare breastfeeding status between Immediate and delayed breastfeeding postpartum contraceptive users by using questionnaire whether each participant is full-breastfeeding, partial-breastfeeding or non-breastfeeding and specify reasons if she's not full-breastfeeding.
Child weight | immediately after contraceptive implant use until 12 weeks after use
  To compare child growth by measuring weight, between Immediate and delayed breastfeeding postpartum contraceptive users.
Child height | immediately after contraceptive implant use until 12 weeks after use
  To compare child growth by measuring height, between Immediate and delayed breastfeeding postpartum contraceptive users.

CONTACTS AND LOCATIONS:
Overall Officials: Unnop Jaisamrarn, M.D., Study Chair — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Derived] Sothornwit J, Kaewrudee S, Lumbiganon P, Pattanittum P, Averbach SH. Immediate versus delayed postpartum insertion of contraceptive implant and IUD for contraception. Cochrane Database Syst Rev. 2022 Oct 27;10(10):CD011913. doi: 10.1002/14651858.CD011913.pub3. PMID 36302159